CLINICAL TRIAL: NCT03177512
Title: LYNX: A Novel Mobile App to Support Linkage to HIV/STI Testing and Pre-exposure Prophylaxis (PrEP) for Young Men Who Have Sex With Men
Brief Title: LYNX: A Novel Mobile App to Support Linkage to HIV/STI Testing PrEP for Young Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: Cook County Health & Hospitals System (Other); Duke University (Other); Emory University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); San Francisco Department of Public Health (Other Government); University of California, San Francisco (Other); University of North Carolina, Chapel Hill (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Albert Liu, Clinical Research Director, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-21876; U19HD089881 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-06-06 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: HIV; Sexually Transmitted Diseases; Risk Reduction; Pre-Exposure Prophylaxis
Keywords: PrEP; HIV Testing; STI Testing; Mobile app; Technology; Young men who have sex with men
MeSH Terms: conditions — Sexually Transmitted Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYNX Mobile App (Experimental)
  Interventions: Behavioral: LYNX Mobile App
- Control (No Intervention): Participants in this study arm will receive local standard of care for linkage to PrEP and HIV/STI testing.

INTERVENTIONS:
Behavioral: LYNX Mobile App — Access to the LYNX mobile app which includes the Sex Pro score tool, PrEP videos, HIV/STI testing reminders and geo-location features.
  Arms: LYNX Mobile App

SUMMARY:
This study is testing the acceptability and feasibility of a highly interactive mobile application (app) to promote HIV/sexually transmitted infection (STI) testing and uptake of pre-exposure prophylaxis (PrEP) among young men who have sex with men (YMSM).

DETAILED DESCRIPTION:
Using the Information-Motivation-Behavior Skills (IMB) model, we have developed LYNX, a highly interactive mobile app to promote accurate risk perception and increase HIV/STI testing and linkage to PrEP among young men who have sex with men (YMSM). Key components of the app include Sex Pro (a personalized HIV risk score), a sex diary to facilitate accurate data collection; HIV/STI testing information and reminders; access to home HIV/STI testing options; a geospatial-based locator of HIV/STI testing sites and PrEP clinics; PrEP information and videos; and online PrEP navigation.

This study is part of the iTech NIH U19, which has an overall goal to develop innovative technology-focused interventions addressing the HIV prevention and care continuum for youth.

ELIGIBILITY:
Inclusion Criteria:

* No HIV test in the past 3 months (self-reported).
* Not known to be HIV-infected (self-reported).
* Not currently taking PrEP (self-reported).
* Owns an Apple operating system (iOS) or Android mobile phone and willing and able to download the LYNX app onto their phone.
* Willing and able to attend an in-person baseline visit in the Tampa or Chicago area.
* Able to understand, read, and speak English.
* Participants ages 15-18: self-report at least one episode of anal intercourse with a male or transfemale partner during the last 6 months
* Participants ages 19-24: self-report evidence of high risk for acquiring HIV infection including at least one of the following:

  1. at least one episode of condomless anal sex with an HIV-positive or unknown HIV status male or transfemale partner during the last 6 months; or
  2. Anal sex with 2 or more male and/or transfemale partners during the last 6 months; or
  3. Exchange of money, gifts, shelter, or drugs for anal sex with a male or transfemale partner during the last 6 months; or
  4. Sex with a male or transfemale partner and has had an STI during the last 6 months.

Exclusion Criteria:

* Currently enrolled in another HIV intervention study
* Prior enrollment in an HIV vaccine trial with receipt of experimental vaccine product
* Enrollment in an earlier phase of LYNX study
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender male
Enrollment: 61 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, M.D., MPH, Study Chair — Bridge HIV, San Francisco Department of Public Health; Hyman Scott, M.D., MPH, Study Chair — Bridge HIV, San Francisco Department of Public Health
Locations (2):
- United States (2):
  - University of South Florida, Department of Pediatrics, Tampa, Florida
  - The CORE Center, Cook County Health and Hospitals System, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu AY, Torres TS, Alleyne CD, Vinson J, Bojan K, Serrano PA, Oyedele T, Garcia A, Enriquez-Bruce E, Emmanuel P, Jones J, Muessig KE, Buchbinder SP, Sullivan P, Hightow-Weidman LB, Scott H. Developing a Novel Mobile App to Support HIV Testing and Pre-Exposure Prophylaxis Uptake Among Men Who Have Sex With Men: Formative and Technical Pilot Study. JMIR Hum Factors. 2025 May 29;12:e62830. doi: 10.2196/62830. PMID 40440084
- [Derived] Liu A, Coleman K, Bojan K, Serrano PA, Oyedele T, Garcia A, Enriquez-Bruce E, Emmanuel P, Jones J, Sullivan P, Hightow-Weidman L, Buchbinder S, Scott H. Developing a Mobile App (LYNX) to Support Linkage to HIV/Sexually Transmitted Infection Testing and Pre-Exposure Prophylaxis for Young Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 25;8(1):e10659. doi: 10.2196/10659. PMID 30681964

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LYNX Mobile App | Control
Started | 40 | 21
Completed | 31 | 18
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYNX Mobile App | Control | Total
Number analyzed (Participants) | 40 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.23 (2.55) | 20.52 (2.73) | 20.33 (2.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 21 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 29 | 14 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3
  Black | 9 | 6 | 15
  White | 20 | 14 | 34
  Other/multiple | 7 | 0 | 7
  Declined to answer | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: System Usability Scale: a validated 10-measure scale that assesses subjective usability of a system, or, in this case, an app. Range of scale is 0-100, with higher scores indicating higher acceptability.
Time Frame: 3 months
Population: Participants in the LYNX Mobile App arm who completed assessment at month 3. Two participants answered "Declined to answer" - SUS was calculated out of 32 complete responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 32 | 0
units on a scale | 75.63 (14.59) |

2. Primary Outcome: Feasibility: Number of Participants Who Opened the App at Least Once by Month 3 Time Point
Description: Opened the app at least once by Month 3 time point
Time Frame: 3 months
Population: Feasibility was only assessed in the intervention arm. One participant was missing from the paradata and not included in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 39 | 0
Participants | 38 |

3. Secondary Outcome: Frequency of App Use
Description: Number of login sessions
Time Frame: 6 months
Population: Frequency of app use was only assessed in the intervention arm. One participant was missing from the paradata and not included in the denominator.
Measure: Mean (Standard Deviation); unit: Number of login sessions
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 39 | 0
Number of login sessions | 15.16 (11.73) |

4. Secondary Outcome: Number of Participants Using Different Parts of the App
Description: Use of each app component based on paradata from the mobile app
Time Frame: 6 months
Population: Analysis only included participants in the intervention arm. One participant was missing from the paradata and not included in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 39 | 0
Participants
  Home page | 38 |
  Diary | 37 |
  Testing | 37 |
  Navigation Chat | 33 |
  Navigation PrEP | 35 |
  SexPro | 34 |
  Activity calendar | 32 |
  Insights | 29 |
  Sex trends | 30 |
  Testing map | 30 |
  Encounter | 29 |
  Profile | 27 |
  PrEP map | 23 |
  Top 5 | 23 |
  Badges | 24 |
  PrEP facts | 12 |
  PrEP videos | 5 |

5. Secondary Outcome: Number of Participants Who Ordered HIV/STI Home Testing Kits, Condoms and Lube
Description: Number of Participants who ordered HIV/STI home testing kits, condom and lube
Time Frame: 6 months
Population: Only includes participants in the intervention arm, as home test kits could only be ordered through the app for participants in the LYNX mobile app arm
Measure: Number; unit: participants
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 40 | 0
participants
  Oraquick testing kit orders | 38 |
  STI testing kit orders | 37 |
  Condom orders | 29 |
  Lube orders | 19 |

6. Secondary Outcome: Number of Participants Reporting HIV Testing Over 6 Months
Description: Self-report HIV testing during 6 month study
Time Frame: 6 months
Population: Participants analyzed included those who had completed at least one follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 35 | 18
Participants | 28 | 11

7. Secondary Outcome: PrEP Uptake as Measured by Self Report
Description: Self-report of PrEP use
Time Frame: 6 months
Population: Participants analyzed included those who completed at least one follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | LYNX Mobile App | Control
Number analyzed (Participants) | 34 | 18
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the 6 month trial
Arm/Group | LYNX Mobile App | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/21
Other Adverse Events (participants affected / at risk) | 0/40 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03177512/Prot_SAP_000.pdf